CLINICAL TRIAL: NCT04927988
Title: Blood Components Changes by Using of Ringer's Lactated as Detergent In Autologous Blood Cell Transfusion: A Prospective, Single-center, Open, and Single-arm Clinical Trial
Brief Title: Blood Components Changes by Using of Ringer's Lactated as Detergent In Autologous Blood Cell Transfusion
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: halted by the pandemic of COVID-19
Sponsor: Maternal and Child Health Hospital of Foshan (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCHHFoshan-2101
Record Dates: First submitted 2021-06-09; First posted 2021-06-16 (Actual); Last update posted 2023-04-25 (Actual); Status verified 2023-04

CONDITIONS: Placenta Accreta Spectrum
Keywords: Placenta Accreta Spectrum; Autologous Blood Cell Transfusion; Blood Components
MeSH Terms: conditions — Placenta Accreta | interventions — Ringer's Lactate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Arm 1. (Other): Using of Ringer's Lactated
  Interventions: Other: Ringer's Lactated

INTERVENTIONS:
Other: Ringer's Lactated — Using of Ringer's Lactated In Autologous Blood Cell Transfusion

SUMMARY:
Placenta accreta spectrum (PAS) disorders are associated with increased maternal morbidity and mortality related to life-threatening hemorrhage, and greater potential need for blood transfusion. Clinical evidences have confirmed that the use of autologous blood cell transfusion is safe and effective for patients with obstetric haemorrhage. Normal saline is the solution recommended for red cell washing, administration and salvage. However, there is growing concern that normal saline is more toxic than balanced, buffered crystalloids such as Lactated Ringer's and Plasma-Lyte. The purpose of this study is to evaluate the blood components using of Ringer's Lactated by a prospective, single-center, open, and single-arm clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* Between 18 and 45 years old
* Without health problem nor disease requiring regular medical treatment

Exclusion Criteria:

* subject with contraindication for drawing blood
* Subject with physical or mental disability or restriction of liberty that would prevent autotransfusion

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2021-10 (Estimated); Primary Completion 2022-09 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Change in hematological parameters | Baseline (Day 1), until 2 days after autotransfusion
  erythrocytes (/µL)
Change in hematological parameters | Baseline (Day 1), until 2 days after autotransfusion
  hemoglobin (g/dL)
Change in hematological parameters | Baseline (Day 1), until 2 days after autotransfusion
  Mean corpuscular volume (fL)

CONTACTS AND LOCATIONS:
Locations (1):
- Maternal and Child Health Hospital of Foshan, Foshan, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided